CLINICAL TRIAL: NCT01751347
Title: Bupivacaine Versus Lidocaine Local Anesthesia in Elective Outpatient Hand Surgery: A Randomized Controlled Trial
Brief Title: Bupivacaine Versus Lidocaine Local Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H12-03477
Record Dates: First submitted 2012-12-13; First posted 2012-12-18 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Carpal Tunnel Syndrome; Trigger Finger
Keywords: Local anesthetics; Elective hand surgeries
MeSH Terms: conditions — Carpal Tunnel Syndrome; Trigger Finger Disorder | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Active Comparator): Subjects randomized to this treatment arm will receive lidocaine during their elective hand surgery.
  Interventions: Drug: Lidocaine
- Bupivacaine (Experimental): Subjects randomized to this treatment arm will receive bupivacaine during their elective hand surgery.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Local anesthetics
  Arms: Bupivacaine
Drug: Lidocaine — Local anesthetics
  Arms: Lidocaine

SUMMARY:
The use of local anesthetics has become an important aspect of pain management in surgical settings and is currently recommended in pain management guidelines.

Elective outpatient hand surgeries, such as carpal tunnel or trigger finger release, cause minimum tissue disruption and are short in duration. As a result, these local anesthetic agents are a major component in post-operative pain control. The most commonly used local anesthetic agents are Lidocaine and Bupivacaine. Lidocaine acts faster (within 2-5 minutes of injection) and for this reason is often favored in outpatient setting for pre-incisional injection. However its effects only last up to 2 hours, without epinephrine, and 3 hours, with epinephrine. On the other hand, Bupivacaine, has a slower onset of action (about 5-10 minutes after injection) but its effects last much longer, for about 4-8 hours. The delay in onset of action makes it a less popular option as a primary source of local anesthesia in outpatient hand surgery.

Given the longer duration of anesthesia offered by Bupivacaine, the investigators believe that by giving it pre-operatively in elective outpatient hand surgeries will offer more effective post operative pain control compared to using Lidocaine only. There is limited published data confirming the effectiveness of use of pre-operative Bupivicaine in improved postoperative pain control and decreased consumption of narcotics. Therefore, the aim in this study is to compare the postoperative pain experienced by patients undergoing either elective carpal tunnel release or trigger finger release as well as their use of pain medications when the incision site is infiltrated preemptively with Lidocaine versus Bupivacaine.

The investigators believe that adequate post surgical pain control is essential for patients' full functional recovery. Poorly controlled post surgical pain increases incidence of surgery related complications and thus increased health care costs. It can also reduce patients' mobility, delay their return to full function,. If poorly controlled, post surgical pain may progress to chronic pain and rarely complex regional pain syndromes may ensue.

DETAILED DESCRIPTION:
Subjects will be randomized to receive either 10ml of 0.5% Bupivacaine with 1:200,000 Epinephrine or 10 ml of 1% Lidocaine with 1:100,000 Epinephrine.

In the case of a single digit surgery such as the trigger finger release, the dose will be adjusted to 5ml of 0.5% Bupivacaine with 1:200,000 Epinephrine or 5ml of 1% Lidocaine with 1:100,000 Epinephrine.

An additional 5ml of study drug will be prepared in a separate syringe and administered when needed.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 90 year old
* Able to provide informed consent
* Consent to participate
* Carpal tunnel release surgery or Trigger finger release surgery
* Single procedure

Exclusion Criteria:

* Unable to consent
* Do not consent to participate
* Known Lidocaine or Bupivacaine allergy
* Known Epinephrine allergy or contra indication
* Known Codeine allergy
* Pregnant
* More than one procedure is being performed at the same setting

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
amount of oral analgesic used post procedure | up to 2 weeks post surgery
  Total amount of oral analgesic a subject uses from the day of surgery to 2 weeks post surgery.

SECONDARY OUTCOMES:
Post operative pain | up to 2 weeks post surgery
  Pain (subject reported pain scores) experienced at injection, during surgical procedure and post operative pain experienced by subject up to 2 weeks post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Brown, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada